CLINICAL TRIAL: NCT01045629
Title: Competence Ability Study in People With Schizophrenia
Acronym: CompSchizo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: IRB TCVGH, Taichung Veterans General Hospital
Other Study IDs: C09080
Record Dates: First submitted 2010-01-06; First posted 2010-01-11 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Schizophrenia; Competence
Keywords: schizophrenia; PANSS
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SchizoComp: Competence Ability of schizophrenia
  Interventions: Other: Consent form education
- NonSchizoComp: Competence of Non-schizophrenia

INTERVENTIONS:
Other: Consent form education — Randomly stratified schizophrenic patients group, some receive consent form education, the others not.
  Groups: SchizoComp

SUMMARY:
The goal of this research is to understand whether schizophrenic patients are capable of comprehending clinical trial consent form or influenced by disease, also after intensified educational illustration for "understanding of consent form", their comprehension increased or not, in order to protect patient's right.

DETAILED DESCRIPTION:
The goal of this research is to understand whether schizophrenic patients are capable of comprehending clinical trial consent form or influenced by disease, also after intensified educational illustration for "understanding of consent form", their comprehension will increase or not, in order to protect patient's right. First week, inform the patient a putative goal and method of clinical trial medicine research, then using Macarthur comprehension evaluation tool-clinical research Ed., evaluate the understanding of all patients for this putative clinical trial research consent form. For experimental group schizophrenic patients, using PANSS score evaluate seriousness of their symptom. 2 weeks later, randomly stratify schizophrenic patients into 2 groups, one give educational intervention for consent form, the other does not, then evaluate again with Macarthur comprehension evaluation tool-clinical research Ed. and PANSS score.

ELIGIBILITY:
Inclusion Criteria:

Experimental group

1. Age between 20 to 60, all genders.
2. Psychiatry doctor diagnosed who met DSMIV-TR criteria schizophrenia.
3. Participants require adequate ability to have a interview about 60-70min (include PANSS and Macarthur comprehension evaluation tool-clinical research Ed.).

Control group

1. Age between 20 to 60, all genders.
2. Psychiatry doctor diagnosed who exclude DSMIV-TR axis. I and II.
3. Participants require adequate ability to have a interview about 30min (include PANSS and Macarthur comprehension evaluation tool-clinical research Ed.).

Exclusion Criteria:

Experimental group and control group

Participants have no adequate ability to have a interview about 60-70min (include PANSS and Macarthur comprehension evaluation tool-clinical research Ed.).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Schizophrenic patients and control; PANSS score; Macarthur comprehension evaluation tool-clinical research Ed.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tsuo-Hung Lan, MD., PhD., Study Director — Taichung Veterans General Hospital; Tsuo-Hung Lan, MD.,PhD, Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan